CLINICAL TRIAL: NCT04275713
Title: Altered Tumor Oxygenation by Metformin, a Potential Step in Overcoming Radiotherapy Resistance in Locally Advanced Cervical Cancer.
Brief Title: Altered Tumor Oxygenation by Metformin, a Potential Step in Overcoming Radiotherapy Resistance in LACC
Acronym: METOXY-LACC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kjersti Bruheim, Principal investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METOXY-LACC
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Metformin; Cisplatin

STUDY DESIGN:
Intervention Model Description: Patients are randomized to intervention Group (metformin in combination with radiotherapy) or standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Chemoradiotherapy +/- metformin (Experimental): Metformin will be given orally at doses of 850 mg twice a day. Metformin will be started one week prior to the start of standard cisplatin-based chemoradiotherapy, and will be continued throughout the entire radiation treatment
  Interventions: Drug: Metformin; Drug: Cisplatin
- Standard chemoradiotherapy (Active Comparator): Standard chemoradiotherapy is given as a combination of EBRT and IGT:
  * 45 Gy in 1.8 Gy/fraction to the pelvis/abdomen, 5 fractions/week
  * 55-57.5 Gy in 2.2-2.3 Gy/fraction to pathological lymph nodes as a simultaneously integrated boost (SIB)
  * 4 fractions of brachytherapy, 7.8 Gy/fraction, to the cervix
  * Concomitant Cisplatin weekly during the external beam radiotherapy (EBRT)
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Metformin — Metformin is an oral antidiabetic drug
  Arms: Standard Chemoradiotherapy +/- metformin
Drug: Cisplatin — Cisplatin 40 mg/m2 given intravenously once a week, maximum 6 cycles

SUMMARY:
Poor tumor oxygenation (hypoxia) is an established negative prognostic and predictive factor in locally advanced cervical cancer (LACC). Hypoxia-modifying measures implemented in the clinic are lacking.

Metformin is a well-known, well-tolerated and low-cost drug used for decades in the treatment of type 2- diabetes. Recent studies suggest an improved tumor oxygenation by metformin potentially improving radiotherapy response and patient outcome.

This study is a randomized, phase II, open label study in patients with LACC where patients are randomized to standard cisplatin-based chemoradiotherapy +/- Metformin.

Metformin will be started one week prior to the start of chemoradiotherapy, and will be continued throughout the entire radiation treatment.

Tumor oxygenation will be evaluated by gene signatures and MRI- parameters.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cervical cancer (squamous cell carcinoma, adenocarcinoma and adenosquamous carcinoma)

  * Planned for radical chemoradiotherapy
  * Over 18 years
  * Speaks and understands Norwegian
  * ECOG 0-1
  * Cervical tumor available for biopsy by gynecological examination
  * Hemoglobin ≥ 9 g/dL (blood transfusions are allowed)
  * Leukocytes ≥ 3,5 x 10^9/L 18
  * Absolute neutrophil count ≥ 1,5 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Total bilirubin ≤ 25 umol/L
  * AST/ALT ≤ 2,5 x institutional upper limit
  * Creatinine ≤ 90 or creatinine clearance ≥ 60 ml/min/1.73m2 Patients with elevated creatinine secondary to hydronephrosis may be eligible if renal function returns to normal after inserting an internal stent or nephrostomy
  * Women of childbearing potential (WOCBP) should have a negative highly sensitive serum pregnancy test within 72 hours prior to receiving the first dose of study medication.

Exclusion Criteria:

* Evidence of distant metastasis. Suspicious paraaortic lymph nodes below the renal vessel are allowed if they are covered by the radiation field
* Patients who have received other cancer treatments for their cervical cancer
* Patients who receive other experimental drugs
* Known diabetes mellitus
* Currently taking Metformin or any other antidiabetic drugs (sulfonylureas, thiazolidinediones, insulin)
* History of allergic reaction attributed to compounds of similar chemical or biologic composition to metformin
* Contraindications such as

  * Hypersensitivity to the active substance or to any of the excipients listed Section 6.1.
  * Severe renal failure (GFR <30 ml / min).
  * Acute conditions leading to the risk of renal impairment, eg: dehydration, severe infectious conditions, shock.
  * Disease that can cause tissue hypoxia (especially acute illness or exacerbation of chronic illness), such as: acute decompensated heart failure, lung failure, recent heart attack, shock.
  * Liver failure, acute alcohol intoxication, alcoholism.
* Any condition associated with increased risk of metformin- induced lactic acidosis (congestive heart failure defined as New York Heart Association (NYHA) class III or IV functional status, history of acidosis of any kind)
* Uncontrolled intercurrent somatic illness including, but not limited to, ongoing or active serious infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction within 6 months and cerebrovascular disease with previous stroke
* Already on medication with increased risk of lactic acidosis
* Patients who are pregnant or breastfeeding are excluded due to risk of teratogenic and abortifacient effects of radiotherapy and cisplatin, and the potential risk of adverse effect of nursing infants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Metformin dependent changes in hypoxia-related gene expression. | baseline and one week
  * A hypoxia related 6-gene expression signature analyzed by RNA-sequencing will be obtained before and after one week of metformin
  * The signature consist of the following six genes: ERO1A, DDIT3, KCTD11, P4HA2, STC2, UPK1A

SECONDARY OUTCOMES:
Metformin dependent changes in MRI-parameters. | baseline and one week
  * Diffusion-weighted MRI and Dynamic Contrast-Enhanced MRI will be obtained before and after one week of metformin.
  * Hypoxic tumor fraction on MRI will be calculated using the combined information from DWI- and DCE-MRI
Metformin dependent change in acute toxicity | baseline, 4 weeks, end of treatment (about 7 weeks), 3 month follow-up
  - Physician-reported acute toxicity will be assessed with validated questionnaires (CTCAE version 3 and 4).
Metformin dependent change in tumor volume during treatment | Baseline and about 4 weeks
  - Tumor volume will be measured on T2W-MRI before the start of treatment and at the first fraction of brachytherapy

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Bruheim, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No